CLINICAL TRIAL: NCT00005674
Title: Clinical Trial of Creatine in Amyotrophic Lateral Sclerosis [ALS]
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Muscular Dystrophy Association (Other)
Purpose: Treatment
Other Study IDs: NCRR-M01RR00036-0745; M01RR000036 (NIH)
Record Dates: First submitted 2000-05-26; First posted 2000-05-29 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Creatine

INTERVENTIONS:
Drug: Creatine

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of creatine treatment in amyotrophic lateral sclerosis (ALS). There is currently no known effective treatment for ALS. It is known that nerve cells die in the brains and spinal cords of patients with ALS but the cause of the cell death is unknown. It has been shown that there is overactive nerve activity due to increased levels of a chemical called glutamate and that there is abnormal cellular metabolism along with increased production of substance called "free radicals." Improving cellular metabolism and readjusting the activity of glutamate in the brain may be beneficial to ALS patients.

Creatine is a naturally occurring compound, which improves energy metabolism in cells. Creatine has been given to patients with energy metabolism defects in their muscles, and to athletes. Creatine improves survival in a mouse model of ALS. Three human subjects with ALS have received creatine for up to six months without any side effects. Overall, creatine has been well tolerated and safe.

DETAILED DESCRIPTION:
Half of the subjects in this study will be selected by chance to receive creatine treatment for 6 months and the other half to receive placebo. Neither the subject nor the investigator will know which drug the subject is receiving, although this information will be available in case of emergency. It is anticipated that all subjects will have the choice to receive creatine after the 6 months study in an open-label study for an additional 12 months. A total of 114 patients will participate at 15 centers. Approximately 8 subjects will be enrolled at the Washington University.

The effectiveness of creatine will be determined first by assessing any changes in strength in the arms and second by changes in grip strength, functional activities, electromyography changes or changes of the level of SOH 2'dG in the urine.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of definite, probably or laboratory supported probably ALS, either sporadic or familial ALS according to a modified El Escorial criteria
* Willing and able to give informed consent
* FVC greater than or equal to 50% predicted
* Evidence of abnormality in upper and/or lower extremity motor function (clinical evidence of muscle atrophy and weakness in an upper and/or lower extremity). The patient should have at least 4 or 8 testable upper extremity muscle groups.
* Subjects may take riluzole. Riluzole must have been at stable doses for at least thirty days prior to baseline visit.
* If woman of childbearing age, must be non-lactating and surgically sterile or using an effective method of birth control (double barrier or oral contraceptive) and have a negative pregnancy test
* Disease duration less than five years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States